CLINICAL TRIAL: NCT03201146
Title: A Phase 1/2 Study of Apatinib in Combination With AP(Pemetrexed/Cisplatin) or AC(Pemetrexed/Carboplatin) as First-line Chemotherapy for Advanced Epidermal Growth Factor Receptor(EGFR) Wild Type Non-squamous Non-small Cell Lung Cancer
Brief Title: Apatinib Combine With Platinum-Based Doublet Chemotherapy for First-line Treatment of Advanced NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, You Lu,MD, MD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009L03464
Record Dates: First submitted 2017-06-25; First posted 2017-06-28 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Combination Chemotherapy; Apatinib
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — apatinib; Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Apatinib 750mg + AP or AC (Experimental): Phase 1 study of Apatinib in combination with platinum-based doublet chemotherapy.
  Interventions: Drug: AP or AC; Drug: Apatinib 750mg
- Apatinib 500mg + AP or AC (Experimental): Phase 1 study of Apatinib in combination with platinum-based doublet chemotherapy.
  Interventions: Drug: AP or AC; Drug: Apatinib 500mg
- Apatinib 250mg + AP or AC (Experimental): Phase 1 study of Apatinib in combination with platinum-based doublet chemotherapy(PBDC).
  Interventions: Drug: AP or AC; Drug: Apatinib 250mg
- Apatinib (Experimental): Phase 2 study of Apatinib in combination with platinum-based doublet chemotherapy(PBDC).
  Interventions: Drug: Apatinib; Drug: AP or AC
- AP or AC (Active Comparator): Pemetrexed/Cisplatin(AP) or Pemetrexed/Carboplatin(AC), The platinum-based doublet chemotherapy, as the control group in the phase 2 study.
  Interventions: Drug: AP or AC

INTERVENTIONS:
Drug: Apatinib — Doses to be determined following the completion of Phase I of the study.
  Other Names: YN968D1
  Arms: Apatinib
Drug: AP or AC — Pemetrexed(A) 500mg/m2, IV, Day 1; Cisplatin(P) 25mg/m2,IV,Day 1-3 or Carboplatin(C) area under curve(AUC)=5, IV, Day 1; AP or AC will be administered every 21 days starting on Day 1.
  Other Names: Pemetrexed/Cisplatin or Pemetrexed/Carboplatin
Drug: Apatinib 250mg — 250mg/d,q.d.,p.o.every 21 days.
  Other Names: YN968D1
  Arms: Apatinib 250mg + AP or AC
Drug: Apatinib 500mg — 500mg/d,q.d.,p.o.every 21 days.
  Other Names: YN968D1
  Arms: Apatinib 500mg + AP or AC
Drug: Apatinib 750mg — 750mg/d,q.d.,p.o.every 21 days.
  Other Names: YN968D1
  Arms: Apatinib 750mg + AP or AC

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of Apatinib in combination with AP(Pemetrexed/Carboplatin) or AC(Pemetrexed/Carboplatin) as first-line chemotherapy in subjects with advanced EGFR wild type non-squamous non-small cell lung cancer(NSCLC).

DETAILED DESCRIPTION:
Apatinib, an oral highly potent tyrosine-kinase inhibitor targeting VEGFR-2, has demonstrated improved survival in previously treated patients with advanced non-small-cell lung cancer(NSCLC).

The phase I study is conducted to explore the safety, tolerability, dose-limiting toxicities(DLT), Maximum Tolerable Dose(MTD), and preliminary anti-tumor activity of Apatinib combined with platinum-based doublet chemotherapy(PB-DC) in first-line advanced EGFR wild type non-squamous non-small cell lung cancer. This will use a dose reduction trial design. A cohort of 3~6 subjects will be enrolled at each dose level, If 0 of 3 or ≤ 1 of 6 subjects experience a DLT, the phase I trial will stop and the current dose will be considered the MTD. If 1 of 6 or more subjects experiences a DLT, dose reduce to the next dose will occur.

Following completion of the dose de-escalation trial and determination of MTD, A randomized controlled trial(RCT) including 30 subjects may be enrolled to further evaluate safety, tolerability, and preliminary anti-tumor activity of Apatinib in combination with platinum-based doublet chemotherapy(PB-DC) in the same target population.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed the informed consent form prior to patient entry.
* 2. ≥ 18 and ≤ 70 years of age.
* 3. Histologically or pathologically confirmed non-squamous EGFR wild-type, ALK-rearrangement negative, stage IV non-small cell lung cancer(NSCLC).
* 4. Must have at least one measurable lesion as per RECIST 1.1 defined as a lesion that is 10mm in longest diameter or lymph node that is 15mm in short axis imaged by CT scan, prior topical treatment, such as radiotherapy or cryosurgery to the lesions is not allowed.
* 5. No prior systemic chemotherapy for advanced or metastatic NSCLC.
* 6. Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
* 7. Life expectancy of more than 3 months.
* 8. Adequate bone marrow function : WBC ≥ 3.0 ×10 E+9/L, neutrophil ≥ 1.5 × 10 E+9/L, platelets ≥ 80 × 10E+9/L,Hb ≥ 10.0g/dL.
* 9. Adequate hepatic and renal functions: a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL), a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis, a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault).
* 10. With normal coagulation function: INR and PTT, each ≤ 1.5 x ULN.
* 11. Adequate cardiovascular function: left ventricular ejection fraction (LVEF) ≥ 50%, QTcF ≤ 450 msec.
* 12. Alkaline phosphatase ≤ 2.5 x ULN.
* 13. The subjects are willing to coordinate with the follow-up with good compliance.
* 14. Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug.

Exclusion Criteria:

* 1. Patients with active brain metastasis, carcinomatous meningitis, or spinal compression, or disease of brain or pia mater according to the screening test, imaging, CT or MRI tests (patients who have completed the treatment and in a stable condition 21 days before screening could be included, but brain MRI, CT or venography is required to confirm that there are no brain hemorrhage symptoms).
* 2. Patients with uncontrollable hypertension (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg, despite optimal drug therapy).
* 3. Patients with with grade Ⅱ myocardial ischemia or myocardial infarction, poor control of arrhythmias (including QTc interval male ≥ 450 ms, female ≥470 ms).
* 4. According to NYHA standard, grade Ⅲ ~ Ⅳ heart failure, or cardiac color Doppler ultrasound examination showed left ventricular ejection fraction (LVEF) <50%.
* 5. Coagulation dysfunction (INR> 1.5, PT> ULN +4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment.
* 6. Patients treated with anticoagulation agents or Vitamin K antagonist such as Warfarin, heparin, or other similar drugs.
* 7. Patients who had obvious hemoptysis within 2 months before screening, or experienced daily hemoptysis with a volume more than half a tea spoon (2.5ml) or above.
* 8. Patients who experienced bleeding symptoms of clinical significance within 3 months before screening, or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc.
* 9. Patients who manifested arterial/venous thrombus events, e.g. cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening.
* 10. Known genetic or acquired bleeding or bleeding tendency (such as hemophilia, blood coagulation dysfunction, thrombocytopenia, and hypersplenism, etc.).
* 11. Patients who have unhealed wounds or fractures for a long time.
* 12. Patients who received major surgical operations or experienced severe traumatic injuries, bone fracture, or ulcers within 4 weeks before screening.
* 13. Patients with obvious factors affecting absorption of oral drugs, such as difficulties in swallowing, chronic diarrhea and intestinal obstruction, etc.
* 14. Occurrence of abdominal fistula, gastrointestinal perforation, or intraperitoneal abscess within 6 months before screening.
* 15. Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g.
* 16. Patients with active hepatitis B virus or hepatitis c virus infection.
* 17. Active infection requiring antimicrobial treatment, such as antibacterial, antifungal, or antiviral therapy.
* 18. Patients with clinical symptoms, or dropsy of serous cavity requiring surgical treatment (including hydrothorax, ascites, and hydropericardium).
* 19. Patients who have a history of psychotropic drug abuse and are unable to break the habit, or who have a psychogeny.
* 20. Patients who have taken part in other drug clinical tests within 4 weeks before screening.
* 21. Prior VEGFR inhibitor treatment.
* 22. Patients who formerly suffered from or currently are complicated with other uncured malignant tumors, except basal cell carcinoma, carcinoma in situ of cervix and superficial bladder cancer that have been cured.
* 23. Patients who received the treatment with potent CYP3A4 inhibitors within 7 days before screening, or potent CYP3A4 inducers within 12 days before being included.
* 24. Pregnant or lactating women, fertile patients who are unwilling or unable to take effective contraceptive measures.
* 25. Conditions determined by investigators to possibly affect the clinical study or determination of the study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-06-27 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Up to 36 months
  To determine ORR of Apatinib in combination with AP or AC in subjects with advanced EGFR wild type non-squamous non-small cell lung cancer. ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 36 months
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
Disease Control Rate (DCR) | Up to 36 months
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
median Overall Survival | Up to 36 months
  median Overall survival is defined as the time in months from the start of protocol treatment until the date of death, or the date of last follow-up if alive. Kaplan-Meier methods will be used to estimate overall survival.
One-year Overall Survival Rate | Up to 36 months
  Kaplan Meier methods were used to estimate the 1-year survival probabilities for time to death from any cause. Estimates of the 1-year (365 day) survival probabilities and corresponding 95% confidence intervals (CI) were presented by treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li J, Zhao X, Chen L, Guo H, Lv F, Jia K, Yv K, Wang F, Li C, Qian J, Zheng C, Zuo Y. Safety and pharmacokinetics of novel selective vascular endothelial growth factor receptor-2 inhibitor YN968D1 in patients with advanced malignancies. BMC Cancer. 2010 Oct 5;10:529. doi: 10.1186/1471-2407-10-529. PMID 20923544